CLINICAL TRIAL: NCT02878954
Title: Exercise in Peripheral Artery Disease - Gender-specific Differences and Unexplored Opportunities in Women: the GrEnADa-project
Brief Title: Exercise in Peripheral Artery Disease
Acronym: GrEnADa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13072016_Grenada
Record Dates: First submitted 2016-08-11; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention (Other): 160 men and women with PAD will be recruited.
  Interventions: Other: No intervention (Observational study); Other: Control session; Other: Exercise session
- Control session (Other): 40 patients (men and women) will complete this session.
  Interventions: Other: Control session
- Exercise session (Other): 40 patients (men and women) will complete this session.
  Interventions: Other: Exercise session

INTERVENTIONS:
Other: No intervention (Observational study) — 160 patients will be recruited to:
  * Fill in questionnaires related to demographic characteristics, severity of disease and physical activity.
  * Perform a six-minute walk test Comparison between men and women will be performed.
  Arms: No intervention
Other: Control session — Out of the 160 participants of the observational study, at least 40 (20 men and 20 women) will be recruited.
  In the control session participants will be seated in resting position for 15 minutes.
  Arms: Control session; No intervention
Other: Exercise session — 40 patients will perform a single maximal exercise test on a treadmill. Speed will be maintained at 3.2 km/h and the grade will be increased with 2% every 2 min following Gardner's protocol.
  Arms: Exercise session; No intervention

SUMMARY:
This research project aims to investigate the gender-based difference in patients with peripheral artery disease. To attend this, this study has two specific objectives:

Objective 1: To identify gender-specific barriers towards exercise and physical activity in patients with peripheral artery disease (PAD).

Objective 2: To evaluate gender-specific differences in functional capacity and cardiovascular function and regulation in patients with PAD at rest, during and following a single session of maximal exercise.

ELIGIBILITY:
Inclusion Criteria:

* Ankle-brachial index (ABI) ≤ 0.9 in one or two legs
* Fontaine stage II of PAD
* Body mass index <35 kg/m2
* Resting systolic blood pressure (BP) <160 mmHg and diastolic BP <105 mmHg
* Ability to walk at least 2min at 3.2 km/h
* Ability to undertake an incremental treadmill test
* Decrease of at least 15% in ABI after a maximal treadmill test
* Not currently engaging in any regular exercise program

Exclusion Criteria:

* Exercise induced signs of myocardial ischemia or complex ventricular arrhythmias
* Cardiovascular autonomic neuropathy
* Use of beta-blocker
* Nondihydropyridine calcium antagonists or insulin and hormone replacement therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Barriers towards exercise assessed by questionnaires in patients with peripheral artery disease. | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
  After completion of the 6-minute walking test, patients will be asked to fill in the following questionnaires: walking impairment questionnaire, walking estimated-limitation calculated by history (WELCH), San Diego Claudication Questionnaire, SF-36 and two questionnaires for personal and environmental barriers to physical activity.
Gender-specific differences in walk capacity in patients with peripheral artery disease | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
  The measurements of this outcome will be performed in a second visit day, separated by at least 48h from visit 1 (outcome 1).
  Patients will perform a maximal exercise test to determine claudication onset distance (m) defined as the distance walked until the patients first reported pain in the leg during the treadmill test and total walk distance (m) defined as the total distance that the patient was able to walk during the test.
Gender-specific differences in functional capacity in patients with peripheral artery disease | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
  Walking economy defined as VO2 measured during the first stage of the treadmill test and functional capacity defined as VO2 peak obtained during the test will be obtained.

SECONDARY OUTCOMES:
Gender-specific differences in physical activity level measured by accelerometer | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
Gender-specific differences in autonomic modulation at rest and after a maximal exercise test | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
  Autonomic modulation: assessed by spectral analysis of heart rate and systolic blood pressure variabilities. Heart rate (electrocardiogram) and beat-by-beat blood pressure (finometer) will be recorded for 10 min at a sample frequency of 500Hz/channel.
Gender-specific differences in vascular function in patients with peripheral artery disease at rest and after a maximal exercise test | Cross-sectional study. This outcome will be measured through study completion, an average of 18 months.
  Blood flow and blood flow response after reactive hyperemia.